CLINICAL TRIAL: NCT07094633
Title: Comparative Effects of Kegel Versus Clamshell Exercises on Low Back Pain in Women With Uterine Fibroids: A Randomized Clinical Trial
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Faisalabad (Other)
Responsible Party: Principal Investigator, Dr Izza Ayub; PT, Dr Izza Ayub; PT, University of Faisalabad
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: TUF/PB/34/1027/34
Record Dates: First submitted 2025-07-23; First posted 2025-07-30 (Actual); Last update posted 2025-07-30 (Actual); Status verified 2025-02

CONDITIONS: Low Back Pain; Uterine Fibroids (UF)
MeSH Terms: conditions — Low Back Pain; Leiomyoma

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Kegel Exercise Group (Experimental)
  Interventions: Procedure: Kegel Exercise Group
- Clamshell Exercise Group (Active Comparator)
  Interventions: Procedure: Clamshell Exercise Group

INTERVENTIONS:
Procedure: Kegel Exercise Group — The patient was positioned in a supine lying position, with the therapist standing beside them for guidance. They were instructed to engage and contract their pelvic floor muscles for 3 to 5 seconds, followed by a relaxation phase of 3 to 5 seconds.
  Arms: Kegel Exercise Group
Procedure: Clamshell Exercise Group — The patient was positioned in a side-lying posture with both knees flexed at 90 degrees. One hand was placed on the hip for stability, while the other supported the head. The therapist, standing nearby, instructed the patient to lift the top knee as high as comfortably possible while keeping the feet together. The position was held for 3 to 5 seconds, after which the knee was slowly lowered back to the starting position.
  Arms: Clamshell Exercise Group

SUMMARY:
Uterine fibroids represent a significant health concern for many women of reproductive age. Common symptoms include a tilted pelvis, heavy menstrual bleeding, and lower back pain (LBP). Nonspecific LBP is particularly prevalent among individuals aged 30 to 50 years, and it is one of the major symptoms experienced by women with uterine fibroids. Exercise therapy has been shown to be an effective approach for managing this condition. In particular, Kegel exercises and Clamshell exercises have emerged as promising options. Kegel exercises primarily focus on strengthening the pelvic floor muscles, while Clamshell exercises target the pelvic region and play a vital role in alleviating LBP. Therefore, the aim of this study was to compare the effects of Kegel exercises and Clamshell exercises in reducing lower back pain in women with uterine fibroids.

ELIGIBILITY:
Inclusion Criteria:

* Age 30-50 years
* Chronic low back pain for the last 6 months
* History of dysmenorrhea
* Able to perform exercise independently
* Not undergoing other treatments for treating LBP
* Informed consent

Exclusion Criteria:

* History of any surgery or trauma in last 3 months
* Polycystic ovary syndrome (PCOS)
* Any neurological issue
* History of any form of cancer
* History of recent abortion in the previous 3 months
* Cardiac or renal diseases that affect the exercise participation of the patient

Ages: 30 Years to 50 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Gender Based: Yes
Enrollment: 30 (Actual)
Dates: Start 2025-02-14 (Actual); Primary Completion 2025-05-30 (Actual); Study Completion 2025-05-30 (Actual)

PRIMARY OUTCOMES:
Back Pain | 4 weeks
  Numeric pain rating scale (NPRS) is a tool used for measuring pain intensity in which individuals rate their pain from 0 to 10. 0 represents no pain while 10 represents the worst pain. It can be used in verbal, visual or written forms.

SECONDARY OUTCOMES:
Functional Disability | 4 weeks
  Oswestry disability index (ODI) is a questionnaire designed to assess disability level in patients with LBP. It consists of 10 sections with 6 questions, each section is scored from 0-5, higher the score greater the disability.

CONTACTS AND LOCATIONS:
Locations (1):
- The University of Faisalabad, Faisalābad, Pakistan